CLINICAL TRIAL: NCT06556914
Title: Effect of Albumin Replacement on Oxygen Delivery in Sepsis Patients
Status: Recruiting | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: albumin do2
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Sepsis; Intensive Care Unit
Keywords: oxygen delivery; Sepsis; albumin deficiency
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group albumin: The effect of albumin replacement on the measurements will be evaluated by calculating the ECHO findings, blood gas parameters and SOFA score of the study patients before and after albumin replacement. Oxygen delivery will be calculated 6 times in total for 3 days and the SOFA score will be calculated 3 times in total once a day.

SUMMARY:
Fluid resuscitation is a critical component of sepsis treatment. Research has shown that intravenous (IV) fluid therapy in sepsis positively impacts cardiac output and thereby oxygen (O2) delivery through a complex interaction of central venous pressure, right atrial pressure, venous resistance, ventricular compliance, cardiac contractility, and systemic vascular resistance. The 2021 sepsis prevention guidelines recommend balanced crystalloids as first-line therapy. However, no studies in the literature have evaluated the effect of albumin on O2 delivery. In our study, the investigators aim to assess the impact of albumin replacement on O2 delivery in sepsis patients in the intensive care unit.

DETAILED DESCRIPTION:
Patients will be admitted from the emergency room, operating room or medical wards. After obtaining written consent from the patients or their guardians, patients who are followed up in the intensive care unit with a diagnosis of sepsis, patients over the age of 18, who are diagnosed with hypo-albuminemia after more than 4 L/day fluid resuscitation and who undergo albumin replacement will be included in the study. Treatment support for sepsis patients will be organized according to international guidelines and our local protocol, with appropriate antibiotic therapy, fluid infusion (Crystalloids 20 mL/Kg), norepinephrine infusion to keep mean arterial pressure (MAP)>65 mmHg, and infection source control. Demographic information of the patients, sepsis cause, systemic diseases, surgical history, Sequential Organ Failure Assessment (SOFA) score, which shows the severity of the disease, Acute Physiology and Chronic Health Evaluation (APACHE II) score, hemodynamic variables, blood gas parameters, complete blood count and blood biochemistry. values, total daily fluid intake and excretion, and daily fluid balance will be recorded.

For patients with a plasma albumin value below 2.5 d/dL who require 4 L or more of crystalloid per day, 20% Albumin (100 mL) will be administered as an intravenous infusion over a minimum of 15 minutes once a day for 3 days.The effect of albumin replacement on the measurements will be evaluated by calculating the ECHO findings, blood gas parameters and SOFA score of the study patients before and after albumin replacement. Oxygen delivery will be calculated 6 times in total for 3 days and the SOFA score will be calculated 3 times in total once a day.

ELIGIBILITY:
Inclusion Criteria:

* Followed up with a diagnosis of sepsis,
* over 18 years old
* Patients who were diagnosed with hypo-albuminemia after more than 4L/day fluid resuscitation and underwent albumin replacement

Exclusion Criteria:

* Consent is not given by the patient or his/her guardian,
* The initial cause of shock was hypovolemic, cardiogenic or obstructive shock.
* Pregnancy or suspected pregnancy
* Peripheral limb or severe organ ischemia with peripheral artery disease
* Cardiac functions cannot be evaluated optimally by transthoracic echocardiography
* Patients who died within the first 24 hours after intensive care admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Arterial oxygen saturation (SaO2), hemoglobin (Hb), partial pressure of oxygen in the arterial blood (PaO2) values will be obtained by blood gas measurements.
  Cardiac output will be calculated from the parasternal long axis window by transthoracic echocardiography and left ventricular outflow tract (LVOT) measurement. LVOT peak velocity measurement (VTI) will be displayed in PulseWave mode through the apical 5-window window. During measurement, the image will be frozen and VTI will be measured from the widest wave.
  The effect of albumin replacement on the measurements will be evaluated by calculating the ECHO findings, blood gas parameters and SOFA score of the study patients before and after albumin replacement.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
oxygen delivery | Up to 1 hour after albumin replacement
  Effect of albumin replacement on oxygen delivery.Arterial oxygen saturation (SaO2), hemoglobin (Hb), partial pressure of oxygen in the arterial blood (PaO2) values will be obtained by blood gas measurements.DO2(oxygen delivery): CO x 10 x (Hbx1,34x SaO2) When oxygen delivery to tissue is calculated according to this formula, normal values are 5 x 10 x 15 x 1,34 x 0.98 =984 ml/dk.

SECONDARY OUTCOMES:
change in SOFA score | Up to 12 hour after albumin replacement
  Effect of albumin replacement on change in SOFA score. By evaluating the Central nervous system, Cardiovascular system, Respiratory system, Coagulation, Liver and Renal function, each organ system receives a score ranging from 0 (normal) to 4 (most abnormal), with a minimum SOFA score of 0 and a maximum SOFA score of 24.

CONTACTS AND LOCATIONS:
Overall Officials: gamze MD ertaş, specialist, Principal Investigator — Samsun University
Locations (1):
- Samsun University, Samsun, Ilkadım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shasthry SM, Kumar M, Khumuckham JS, Sarin SK. Changes in cardiac output and incidence of volume overload in cirrhotics receiving 20% albumin infusion. Liver Int. 2017 Aug;37(8):1167-1176. doi: 10.1111/liv.13375. Epub 2017 Mar 5. PMID 28135785